CLINICAL TRIAL: NCT02666235
Title: A Randomised Controlled Trial of the Effect of Remote Ischaemic Conditioning on Coronary Endothelial Function in Patients with Angina.
Brief Title: Remote Ischaemic Conditioning and Coronary Endothelial Function (RIC-COR)
Acronym: RIC-COR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: University of Glasgow (Other); Chest, Heart and Stroke Association Scotland (Other); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Principal Investigator, Colin Berry, Professor of Cardiology and Imaging, NHS National Waiting Times Centre Board
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 11/CARD/03; R11/A136 (Other Grant/Funding Number: Chest Heart & Stroke Scotland); 10/S0704/52 (Other: West of Scotland Research Ethics Service)
Record Dates: First submitted 2015-12-24; First posted 2016-01-28 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Preconditioning; Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischaemic conditioning (Active Comparator): Intermittent inflation of a forearm blood pressure cuff for 5 minute periods at 200 mmHg separated by a 5 minute rest interval, repeated successively on 4 occasions over a 40 minute period. The intervention will take place on the ward with the patient obscured from the clinical team by a curtain.
  Interventions: Procedure: Remote ischaemic conditioning
- Control group (Sham Comparator): Sham intervention: Arm cuff placement but without inflation during a 40 minute period. A curtain will obscure the patient from the clinical team during this time. Arm cuff placement, no inflation.
  Interventions: Procedure: Arm cuff placement, no inflation;

INTERVENTIONS:
Procedure: Remote ischaemic conditioning — Intermittent inflation of an arm blood pressure cuff for 5 minute periods at 200 mmHg separated by a 5 minute rest interval, repeated successively on 4 occasions over a 40 minute period. The intervention will take place on the ward with the patient obscured from the clinical team by a drawn curtain. The clinical team and researchers will be masked to the intervention type.
  Other Names: Ischaemic preconditioning; Remote ischemic preconditioning
  Arms: Remote ischaemic conditioning
Procedure: Arm cuff placement, no inflation; — Sham procedure involving arm cuff placement, no inflation: A blood pressure cuff will be placed on the arm for 40 minutes. The cuff will not be inflated. The patient will be in bed behind a curtain on the cardiology ward. The curtain will obscure the patient from the attending cardiology team. The clinical team and researchers will be masked to the intervention type.
  Other Names: Sham procedure
  Arms: Control group

SUMMARY:
Intermittent arm cuff inflation reduces the extent of heart muscle injury at the time of cardiovascular injury. The intervention is known as remote ischaemic conditioning (RIC) however the mechanisms by which RIC acts are incompletely understood.

One mechanism that might explain the benefits of RIC is an improvement in coronary artery function which in turn might help improve blood flow to heart muscle.

The investigators will perform a randomised controlled study of RIC in a minimum of 60 patients with known or suspected angina and in whom coronary angiography with angioplasty would be considered.

Following informed consent before the invasive procedure, the patient will be randomly assigned to the intervention group (cuff inflation protocol) or the control group (cuff placement, no inflation; sham protocol). Following initial coronary angiography, endothelial function will be assessed by intra-coronary infusion of acetylcholine in incremental doses. Coronary diameter will be measured after the procedure using quantitative coronary angiography, by a trained observer blinded to the allocated group. Since a neuro-hormonal response may potentially mediate RIC, a blood test will be performed before and after cuff placement in all patients (active and control groups) to measure circulating molecules known to regulate blood vessel function which may be implicated in a RIC-mediated effect on coronary artery tone.

This study may provide clinically relevant insights into the mechanisms of action of RIC in patients with coronary heart disease.

DETAILED DESCRIPTION:
Intermittent arm cuff inflation reduces the extent of heart muscle injury at the time of cardiovascular injury. The intervention is known as remote ischaemic conditioning (RIC) however the mechanisms by which RIC acts are incompletely understood. One mechanism that might explain the benefits of RIC is an improvement in coronary artery function which in turn might help improve blood flow to heart muscle.

The primary aim is to determine whether intermittent inflation of a blood pressure cuff for 5 min periods at 200 mmHg on 4 occasions separated by 5 minute intervals can improve coronary vascular function compared to cuff placement with no cuff inflation. A secondary aim is to determine whether or not RIC alters the circulating concentrations of small molecules and hormones in systemic blood that regulate coronary endothelial function.

The investigators will perform a randomised controlled trial of RIC in a minimum of 60 patients with known or suspected angina and in whom coronary angiography with angioplasty would be considered. A screening log will be prospectively recorded. In order to be enrolled prior knowledge of the coronary anatomy and disease is necessary, and this information can be obtained by screening referrals for invasive angiography following non-invasive CT coronary angiography, or staged invasive management when angioplasty is intended following initial invasive angiography.

The protocol had initially involved two coronary angiograms with coronary reactivity testing on the same day, with the first angiogram taking place before the RIC-COR intervention and the second angiogram taking place immediately afterwards. However, after enrolling 10 participants it was evident that the total procedure time and hospital stay was unduly long and impractical. Therefore, following consultation with the trial biostatistician, funder and ethics committee, the protocol was amended and the initial angiogram was removed (May 2012). There were no other changes to the study design. Following a change in service arrangements for elective referrals for coronary angioplasty in our hospital, and constraints around staff illness and availability, recruitment was temporarily suspended on logistical grounds (September 2013 to November 2014).

Following informed consent before the invasive procedure, the patient will be randomly assigned to the intervention group (cuff inflation protocol) or the control group (cuff placement, no inflation; sham protocol). The clinical team will be blind to treatment group assignment.

Clinically-indicated coronary angiography will be performed first, including administration of glyceryl trinitrate (200 - 400 micrograms; short acting preparation) to attenuate coronary artery tone. Based on the angiographic findings, the cardiologist will select a coronary artery with minimal or no evidence of coronary artery disease.

Endothelial function will then be assessed in this artery by intra-coronary infusion of acetylcholine (ACh) in incremental doses. Non-endothelium dependent vasodilation will be assessed using intra-coronary administration of glyceryl trinitrate at the end of the infusion protocol.

An infusion catheter will be used to selectively instrument the coronary artery of interest. The factors that influence the selection of a coronary artery for study include 1) minimal or no angiographic evidence of coronary disease, 2) practical considerations for insertion of an intra-coronary catheter ie. vessel tortuosity, calibre. The coronary reactivity protocol involves intra-coronary administration of study drug at a rate of 2 ml/min for 2 minutes in the following order: 1) 0.9% normal saline; 2) ACh 10-6 Molar (M), 3) ACh 10-5M, 4) ACh 10-4M, 5) 0.9% normal saline; and finally, 6) bolus intra-coronary administration of 200-400 micrograms of glyceryl trinitrate. The patient's clinical response will be assessed prospectively, including with continuous haemodynamic recording (heart rate, rhythm, conduction and aortic blood pressure). A 12-lead electrocardiogram (ECG) and cine coronary angiogram will be obtained synchronously at baseline, at the end of each 2 minute infusion, and following nitrate administration.

Coronary diameter will be measured after the procedure using computer-assisted quantitative coronary analysis (QCA) with custom software (eg Medis, Leiden, Netherlands), by a trained observer blinded to the allocated group. The coronary segment for analysis will be located distal to the infusion catheter in the proximal - mid segment of the right coronary artery or a main branch of the left coronary artery. The segment will have minimal or no angiographic evidence of coronary disease. The length of the segment will be 30 mm. The same angiographic projection will be used for all of the analyses. The software will be calibrated on the catheter. Mean lumen diameter and mean coronary area will be computed.

Epicardial spasm, defined as >90% reduction in coronary artery diameter with ischaemic ST-segment changes on the ECG, and microvascular spasm, defined as ischaemic ST-segment changes without epicardial coronary vasoconstriction >90% will be assessed.

ECG changes, including alterations in atrio-ventricular conduction and ST-segment deviation, will be prospectively recorded.

Since a neuro-hormonal response may potentially mediate RIC, a blood test will be performed before and after cuff placement in all patients (active and control groups) to measure circulating molecules known to regulate blood vessel function.

The study data will be analysed by a biostatistician who is independent of the research team.

If the investigators can discover the effects, if any, of RIC on coronary vascular function, then potentially this information would provide new insights into the mechanisms of action of RIC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or over
2. Known or suspected coronary artery disease
3. A clinical indication for coronary angiography.

Exclusion Criteria:

1. Myocardial infarction within 2 weeks
2. History of coronary artery bypass surgery
3. Second or third degree atrioventricular block
4. Written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Coronary artery diameter change | Intra-procedure
  The net percentage change in mean coronary artery diameter (endothelial function) following intra-coronary administration of study drug (ACh or glyceryl trinitrate) compared to baseline.

SECONDARY OUTCOMES:
Circulating molecules reflecting endothelial function and oxidative stress | Peri-procedure; from baseline up to 2 hours
  Circulating concentrations of small molecules and hormones that are mediators of endothelial function and vascular tone.
Mean percentage change in coronary lumen diameter (delta CAD) | Intra-procedure - After intracoronary infusion of intra-coronary acetylcholine
  The investigators aim to assess the percentage change from baseline in mean coronary lumen diameter, if any, in response to graded doses (10-6M, 10-5M, 10-4M) of intra-coronary acetylcholine infusion with each dose administered over a 2 minute period.
Mean percentage coronary vasoconstriction | Intra-procedure - After intracoronary infusion of intra-coronary acetylcholine
  The investigators aim to assess the vasoconstrictor response, if any, to graded doses (10-6M, 10-5M, 10-4M) of intra-coronary acetylcholine infusion with each dose administered over a 2 minute period.
Coronary endothelial dysfunction | Intra-procedure - After intracoronary infusion of intra-coronary acetylcholine
  A decrease in luminal diameter of >20% after intracoronary infusion of acetylcholine.
Mean percentage change in coronary lumen diameter (delta CAD) | Intra-procedure - After intracoronary injection of glyceryl trinitrate
  The investigators aim to assess the percentage change from baseline in mean coronary lumen diameter, if any, following intracoronary injection of glyceryl trinitrate (200-400 micrograms)
Mean percentage coronary vasodilatation | Intra-procedure - After intracoronary injection of glyceryl trinitrate
  The investigators aim to assess the percentage change from baseline in mean coronary lumen diameter, if any, following intracoronary injection of glyceryl trinitrate(200-400 micrograms)
Epicardial coronary artery spasm | Intra-procedure - During intra-coronary infusion of acetylcholine
  Epicardial coronary artery spasm is defined as a reduction in coronary diameter >90% following intracoronary acetylcholine in comparison with baseline resting condition following intracoronary glyceryl trinitrate administration in any epicardial coronary artery segment together with symptoms and ST segment deviation on the ECG. Epicardial artery spasm may be focal or diffuse. Focal constriction was defined as a circumscribed transient vessel narrowing within the borders of 1 isolated or 2 neighbouring coronary segments. Diffuse constriction was diagnosed when the vessel narrowing was observed in ≥2 adjacent coronary segments. Proximal spasm was defined as vasoconstriction occurring in segments 1, 5, 6, or 11. Mid-vessel spasm was recorded when occurring in segments 2, 3, or 7, whereas distal spasm was defined as that occurring in segments 4, 8, 9, 10, 12, 13, 14, or 15. This approach is in line with the guideline recommendations by COVADIS (Eur Heart J 2015; PMID: 26245334).
Microvascular spasm | Intra-procedure - During intra-coronary infusion of acetylcholine
  Microvascular spasm was diagnosed when angina occurred with typical ischaemic ST-segment changes in the absence of epicardial coronary constriction >90% diameter reduction.
ST-segment deviation | Intra-procedure - During intra-coronary infusion of acetylcholine
  ST-segment deviation from the iso-electric line due to ST-segment elevation or ST-segment depression, is a manifestation of myocardial ischaemia. Since remote ischaemic conditioning is postulated to mitigate myocardial ischaemia, the presence and extent of ST-segment deviation will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, PhD FRCP, Principal Investigator — Golden Jubilee National Hospital
Locations (1):
- Golden Jubilee National Hospital, Glasgow, Dunbartonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no data sharing plan, but we have no objection

REFERENCES:
- [Background] Corcoran D, Young R, Cialdella P, McCartney P, Bajrangee A, Hennigan B, Collison D, Carrick D, Shaukat A, Good R, Watkins S, McEntegart M, Watt J, Welsh P, Sattar N, McConnachie A, Oldroyd KG, Berry C. The effects of remote ischaemic preconditioning on coronary artery function in patients with stable coronary artery disease. Int J Cardiol. 2018 Feb 1;252:24-30. doi: 10.1016/j.ijcard.2017.10.082. PMID 29249435
- [Background] Mohri M, Koyanagi M, Egashira K, Tagawa H, Ichiki T, Shimokawa H, Takeshita A. Angina pectoris caused by coronary microvascular spasm. Lancet. 1998 Apr 18;351(9110):1165-9. doi: 10.1016/S0140-6736(97)07329-7. PMID 9643687
- [Background] Cannon RO 3rd, Epstein SE. "Microvascular angina" as a cause of chest pain with angiographically normal coronary arteries. Am J Cardiol. 1988 Jun 1;61(15):1338-43. doi: 10.1016/0002-9149(88)91180-0. No abstract available. PMID 3287885
- [Background] Wei J, Mehta PK, Johnson BD, Samuels B, Kar S, Anderson RD, Azarbal B, Petersen J, Sharaf B, Handberg E, Shufelt C, Kothawade K, Sopko G, Lerman A, Shaw L, Kelsey SF, Pepine CJ, Merz CN. Safety of coronary reactivity testing in women with no obstructive coronary artery disease: results from the NHLBI-sponsored WISE (Women's Ischemia Syndrome Evaluation) study. JACC Cardiovasc Interv. 2012 Jun;5(6):646-53. doi: 10.1016/j.jcin.2012.01.023. PMID 22721660
- [Background] Sato K, Kaikita K, Nakayama N, Horio E, Yoshimura H, Ono T, Ohba K, Tsujita K, Kojima S, Tayama S, Hokimoto S, Matsui K, Sugiyama S, Yamabe H, Ogawa H. Coronary vasomotor response to intracoronary acetylcholine injection, clinical features, and long-term prognosis in 873 consecutive patients with coronary spasm: analysis of a single-center study over 20 years. J Am Heart Assoc. 2013 Jul 15;2(4):e000227. doi: 10.1161/JAHA.113.000227. PMID 23858100
- [Background] Ong P, Athanasiadis A, Borgulya G, Vokshi I, Bastiaenen R, Kubik S, Hill S, Schaufele T, Mahrholdt H, Kaski JC, Sechtem U. Clinical usefulness, angiographic characteristics, and safety evaluation of intracoronary acetylcholine provocation testing among 921 consecutive white patients with unobstructed coronary arteries. Circulation. 2014 Apr 29;129(17):1723-30. doi: 10.1161/CIRCULATIONAHA.113.004096. Epub 2014 Feb 26. PMID 24573349
- [Background] Sara JD, Widmer RJ, Matsuzawa Y, Lennon RJ, Lerman LO, Lerman A. Prevalence of Coronary Microvascular Dysfunction Among Patients With Chest Pain and Nonobstructive Coronary Artery Disease. JACC Cardiovasc Interv. 2015 Sep;8(11):1445-1453. doi: 10.1016/j.jcin.2015.06.017. PMID 26404197
- [Background] Ong P, Athanasiadis A, Borgulya G, Mahrholdt H, Kaski JC, Sechtem U. High prevalence of a pathological response to acetylcholine testing in patients with stable angina pectoris and unobstructed coronary arteries. The ACOVA Study (Abnormal COronary VAsomotion in patients with stable angina and unobstructed coronary arteries). J Am Coll Cardiol. 2012 Feb 14;59(7):655-62. doi: 10.1016/j.jacc.2011.11.015. PMID 22322081
- [Background] Pries AR, Badimon L, Bugiardini R, Camici PG, Dorobantu M, Duncker DJ, Escaned J, Koller A, Piek JJ, de Wit C. Coronary vascular regulation, remodelling, and collateralization: mechanisms and clinical implications on behalf of the working group on coronary pathophysiology and microcirculation. Eur Heart J. 2015 Dec 1;36(45):3134-46. doi: 10.1093/eurheartj/ehv100. Epub 2015 Jun 25. No abstract available. PMID 26112888
- [Background] Pickard JM, Botker HE, Crimi G, Davidson B, Davidson SM, Dutka D, Ferdinandy P, Ganske R, Garcia-Dorado D, Giricz Z, Gourine AV, Heusch G, Kharbanda R, Kleinbongard P, MacAllister R, McIntyre C, Meybohm P, Prunier F, Redington A, Robertson NJ, Suleiman MS, Vanezis A, Walsh S, Yellon DM, Hausenloy DJ. Remote ischemic conditioning: from experimental observation to clinical application: report from the 8th Biennial Hatter Cardiovascular Institute Workshop. Basic Res Cardiol. 2015 Jan;110(1):453. doi: 10.1007/s00395-014-0453-6. Epub 2014 Dec 2. PMID 25449895
- [Background] Hausenloy DJ, Yellon DM. The therapeutic potential of ischemic conditioning: an update. Nat Rev Cardiol. 2011 Jun 21;8(11):619-29. doi: 10.1038/nrcardio.2011.85. PMID 21691310
- [Background] Przyklenk K, Bauer B, Ovize M, Kloner RA, Whittaker P. Regional ischemic 'preconditioning' protects remote virgin myocardium from subsequent sustained coronary occlusion. Circulation. 1993 Mar;87(3):893-9. doi: 10.1161/01.cir.87.3.893. PMID 7680290
- [Background] Loukogeorgakis SP, Williams R, Panagiotidou AT, Kolvekar SK, Donald A, Cole TJ, Yellon DM, Deanfield JE, MacAllister RJ. Transient limb ischemia induces remote preconditioning and remote postconditioning in humans by a K(ATP)-channel dependent mechanism. Circulation. 2007 Sep 18;116(12):1386-95. doi: 10.1161/CIRCULATIONAHA.106.653782. Epub 2007 Aug 27. PMID 17724264
- [Background] Loukogeorgakis SP, Panagiotidou AT, Broadhead MW, Donald A, Deanfield JE, MacAllister RJ. Remote ischemic preconditioning provides early and late protection against endothelial ischemia-reperfusion injury in humans: role of the autonomic nervous system. J Am Coll Cardiol. 2005 Aug 2;46(3):450-6. doi: 10.1016/j.jacc.2005.04.044. PMID 16053957
- [Background] Steensrud T, Li J, Dai X, Manlhiot C, Kharbanda RK, Tropak M, Redington A. Pretreatment with the nitric oxide donor SNAP or nerve transection blocks humoral preconditioning by remote limb ischemia or intra-arterial adenosine. Am J Physiol Heart Circ Physiol. 2010 Nov;299(5):H1598-603. doi: 10.1152/ajpheart.00396.2010. Epub 2010 Aug 27. PMID 20802131
- [Background] Wolfrum S, Schneider K, Heidbreder M, Nienstedt J, Dominiak P, Dendorfer A. Remote preconditioning protects the heart by activating myocardial PKCepsilon-isoform. Cardiovasc Res. 2002 Aug 15;55(3):583-9. doi: 10.1016/s0008-6363(02)00408-x. PMID 12160956
- [Background] Li J, Rohailla S, Gelber N, Rutka J, Sabah N, Gladstone RA, Wei C, Hu P, Kharbanda RK, Redington AN. MicroRNA-144 is a circulating effector of remote ischemic preconditioning. Basic Res Cardiol. 2014;109(5):423. doi: 10.1007/s00395-014-0423-z. Epub 2014 Jul 25. PMID 25060662
- [Background] Jensen RV, Stottrup NB, Kristiansen SB, Botker HE. Release of a humoral circulating cardioprotective factor by remote ischemic preconditioning is dependent on preserved neural pathways in diabetic patients. Basic Res Cardiol. 2012 Sep;107(5):285. doi: 10.1007/s00395-012-0285-1. Epub 2012 Jul 22. PMID 22821347
- [Background] Rassaf T, Totzeck M, Hendgen-Cotta UB, Shiva S, Heusch G, Kelm M. Circulating nitrite contributes to cardioprotection by remote ischemic preconditioning. Circ Res. 2014 May 9;114(10):1601-10. doi: 10.1161/CIRCRESAHA.114.303822. Epub 2014 Mar 18. PMID 24643960
- [Background] Redington KL, Disenhouse T, Strantzas SC, Gladstone R, Wei C, Tropak MB, Dai X, Manlhiot C, Li J, Redington AN. Remote cardioprotection by direct peripheral nerve stimulation and topical capsaicin is mediated by circulating humoral factors. Basic Res Cardiol. 2012 Mar;107(2):241. doi: 10.1007/s00395-011-0241-5. Epub 2012 Jan 10. PMID 22231674
- [Background] Lee BK, Lim HS, Fearon WF, Yong AS, Yamada R, Tanaka S, Lee DP, Yeung AC, Tremmel JA. Invasive evaluation of patients with angina in the absence of obstructive coronary artery disease. Circulation. 2015 Mar 24;131(12):1054-60. doi: 10.1161/CIRCULATIONAHA.114.012636. Epub 2015 Feb 20. PMID 25712205